CLINICAL TRIAL: NCT00254241
Title: Safety and Efficacy of Seroquel in First Episode Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BU-5077-0011
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Last update posted 2009-06-11 (Estimated); Status verified 2009-06

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate; Risperidone

INTERVENTIONS:
Drug: Seroquel and Risperidone

SUMMARY:
To compare the safety, tolerability and efficacy of Seroquel and risperidone in first episode schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35 years Meet ICD-10 criteria for schizophrenia No abnormaility on clinical examination No previous episode of psychosis No previous antipsychotics of any kind in last 3 months

Exclusion Criteria:

* Have received a course of antipsychotics drug treatment prior to entry which may introduce risk factors or interfere with study procedures Have received anticholinergics within 10 days of baseline aseessment Have received mood stabilizers or anti depressants within 2 weeks

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80
Dates: Start 2002-05; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
The proportion of patients developing clinically significant EPS at any point between baseline (day 1) and final assessment

SECONDARY OUTCOMES:
CGI severity of illness
CGI global improvement
PANSS total score and subscales)
Abnormal Involuntary Movement Scale (AIMS)
Dose of anti cholinergic medication
Serum prolactin levels
Proportion of patients discontinuing treatment due to reasons of lack of efficacy or adverse effects
Proportion of patients experiencing relapse.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZenenca
Locations (1):
- Research Site, London, United Kingdom